CLINICAL TRIAL: NCT03015974
Title: Registry of IgA Nephropathy in Chinese Children
Acronym: RACC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: Nanjing PLA General Hospital (Other); Beijing Children's Hospital (Other); Central South University (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Tongji Hospital (Other); Hunan Children's Hospital (Other Government); Shanghai Children's Hospital (Other); Nanjing Children's Hospital (Other); Children's Hospital of Chongqing Medical University (Other); Shandong Provincial Hospital (Other Government); Fuzhou General Hospital (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Children's Hospital of Hebei Province (Other); Guangzhou Women and Children's Medical Center (Other); Jiangxi Province Children's Hospital (Other); Guangzhou First People's Hospital (Other); Xian Children's Hospital (Other Government); Capital Institute of Pediatrics, China (Other); The First Hospital of Jilin University (Other); Wuhan Women and Children's Medical Center (Other); Tianjin Children's Hospital (Other); Chengdu Women's and Children's Central Hospital (Other); The First People's Hospital of Yunnan (Other)
Responsible Party: Principal Investigator, Jie Ding, Prof., Peking University First Hospital
Other Study IDs: 2015[992]
Record Dates: First submitted 2017-01-03; First posted 2017-01-10 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: IgA Nephropathy; Proteinuria in Nephrotic Range; Immunosuppressive Treatment
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Adrenal Cortex Hormones; Steroids; Prednisone; Prednisolone; deflazacort; Cyclophosphamide; Mycophenolic Acid; Dipyridamole; Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — The urine, serum and DNA of participants are expected to be collected and preserved.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- corticosteroid: pediatric IgA nephropathy treated with only corticosteroid
  Interventions: Drug: Corticosteroid; Drug: Dipyridamole; Drug: ACE Inhibitor or Angiotensin receptor antagonist
- corticosteroid and cyclophosphamide: pediatric IgA nephropathy treated with corticosteroid and cyclophosphamide
  Interventions: Drug: Corticosteroid; Drug: Cyclophosphamide; Drug: Dipyridamole; Drug: ACE Inhibitor or Angiotensin receptor antagonist
- corticosteroid and mycophenolate mofetil: pediatric IgA nephropathy treated with corticosteroid and mycophenolate mofetil
  Interventions: Drug: Corticosteroid; Drug: Mycophenolate mofetil; Drug: Dipyridamole; Drug: ACE Inhibitor or Angiotensin receptor antagonist

INTERVENTIONS:
Drug: Corticosteroid
  Other Names: Steroid; Prednisone; Methylprednisone; Prednisolone; Deflazacort
Drug: Cyclophosphamide
  Other Names: CTX
  Groups: corticosteroid and cyclophosphamide
Drug: Mycophenolate mofetil
  Other Names: MMF
  Groups: corticosteroid and mycophenolate mofetil
Drug: Dipyridamole
Drug: ACE Inhibitor or Angiotensin receptor antagonist

SUMMARY:
This study tries to identify the safe and effective treatment option for IgA nephropathy in children. Investigators will perform prospective registration study among 25 pediatric nephrology medical centers in China.

DETAILED DESCRIPTION:
A total of 1200 patients diagnosed as primary IgA nephropathy with nephrotic proteinuria will be enrolled among 25 pediatric nephrology medical centers nationwide, according to the following protocol.

1. Establishment of registration database online.
2. Participants will be enrolled according to the inclusion criteria and exclusion criteria.
3. The following data will be collected prospectively, including demographic data, clinical symptoms, physical examination, laboratory examination, renal pathology, treatment protocol and follow-up.
4. SPSS software (version 14.0; SPSS, Inc., Chicago, IL, USA) will be used for statistical analysis. P value less than 0.05 will be considered significant.

ELIGIBILITY:
In-patients will be enrolled with the following criteria.

Inclusion Criteria:

* Clinical diagnosis of primary IgA nephropathy.
* Presenting with nephrotic proteinuria, defined as 24-hour urinary protein>50mg/kg, or UPC>2.0 mg/mg.
* Informed consent must be signed.

Exclusion Criteria:

* Diagnosed as secondary renal diseases, including lupus nephritis, purpura nephritis, hepatitis B virus associated nephritis, etc.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of 1200 patients diagnosed as primary IgA nephropathy with nephrotic proteinuria will be enrolled among 25 pediatric nephrology medical centers nationwide.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2016-01; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of proteinuria | Two years
  Complete remission is defined as 24-hour urine protein<150mg or UPC<0.3 g/g with normal kidney function. Partial remission is defined as urine protein decreased by more than 50% with normal renal function.
Renal dysfunction | Two years
  Renal dysfunction is defined as eGFR declined by more than 50%.
Hypertension | Two years
  Hypertension is defined as blood pressure higher than age-specific average level. Use of antihypertensive drugs will be recorded.

SECONDARY OUTCOMES:
End stage renal disease(ESRD) | Two years
  ESRD is defined as eGFR<15ml/min/1.73m2, initiation of long-term dialysis or kidney transplant.
Mortality | Two years
  Death of participants will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Ding, Prof., Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided